CLINICAL TRIAL: NCT02091908
Title: Phase III, Stratified, Randomized, Controlled, Observer-Blind, Multicenter Study to Evaluate the Safety, Tolerability, and Immunogenicity of Two Doses of aH5N1 When Administered to Adult and Elderly Subjects With and Without Underlying Medical Conditions.
Brief Title: Safety and Immunogenicity of Two Doses of aH5N1 Vaccine in Adult and Elderly Subjects With and Without Underlying Medical Conditions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V87_25
Record Dates: First submitted 2014-03-07; First posted 2014-03-19 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Influenza, Human
Keywords: Influenza; H5N1; aH5N1; H5N1 vaccine; Pandemic Influenza vaccine; MF59, Adjuvant, Avian flu; Underlying medical conditions; Underlying cardiovascular medical condition; Pandemic vaccine; Charlson Comorbidity Index (CCI); Adjuvanted vaccine
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1: aH5N1 adult (Experimental): aH5N1 healthy and non-healthy adults
  Interventions: Biological: Novartis Investigational H5N1 vaccine
- Arm 2: aH5N1 elderly (Experimental): aH5N1 healthy and non-healthy elderly
  Interventions: Biological: Novartis Investigational H5N1 vaccine
- Arm 3: aTIV adult (Active Comparator): aTIV healthy and non-healthy adults
  Interventions: Biological: Novartis Seasonal Influenza Vaccine
- Arm 4: aTIV elderly (Active Comparator): aTIV healthy and non-healthy elderly
  Interventions: Biological: Novartis Seasonal Influenza Vaccine

INTERVENTIONS:
Biological: Novartis Investigational H5N1 vaccine — 2 doses of 0.5 ml, 3 weeks apart
  Arms: Arm 1: aH5N1 adult
Biological: Novartis Investigational H5N1 vaccine — 2 doses of 0.5 ml, 3 weeks apart
  Arms: Arm 2: aH5N1 elderly
Biological: Novartis Seasonal Influenza Vaccine — 2 doses of 0.5 ml, 3 weeks apart
  Arms: Arm 3: aTIV adult
Biological: Novartis Seasonal Influenza Vaccine — 2 doses of 0.5 ml, 3 weeks apart
  Arms: Arm 4: aTIV elderly

SUMMARY:
Evaluate the safety, immune response and reactogenicity of aH5N1 vaccination in adult (18 through 60 years of age) and elderly (≥61 years of age) subjects with and without underlying medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* - Male and female individuals 18 years of age and older at the time of enrollment who are mentally competent, willing and able to understand the nature and risks of the proposed study, and able to sign the consent form prior to study entry;
* Individuals who are able to comply with all study procedures and requirements;
* Healthy volunteers and volunteers specifically with underlying COPD, cardiovascular disease, diabetes mellitus, peripheral vascular disease, or renal impairment may be eligible;
* Please contact the site for additional eligibility criteria.

Exclusion Criteria:

* Individuals who are not able to follow all the required study procedures for the whole period of the study;
* Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the Investigator, may interfere with the subject's ability to participate in the study;
* Please contact the site for additional eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving seroconversion | day 43
  Seroconversion is defined as hemagglutination inhibition (HI) ≥1:40 for subjects who were seronegative at baseline [day 1 HI titer <1:10] or a minimum 4-fold increase in HI titer for subjects who were seropositive at baseline [day 1 HI titer ≥1:10])
Geometric mean ratios (GMRs) as determined by HI assay | day 43
Percentage of subjects with an HI titer ≥1:40 | day 43
Solicited and unsolicited adverse events | day 202
  In pooled age groups 18 years of age and older subjects who are healthy or with underlying medical condition who have received aTIV or aH5N1 vaccine.

SECONDARY OUTCOMES:
Geometric mean titers (GMTs) as determined by HI | day 1
  HI assay: homologous antibody responses to aH5N1 vaccine 3 weeks after first vaccination (day 22) according to CHMP immunogenicity criteria in adult and elderly subjects who are healthy or with underlying medical condition
Geometric mean ratios (GMRs) as determined by SRH | day 22
Percentage of subjects with an HI titer ≥1:40 | day 22
Percentage of subjects achieving seroconversion | day 22
  Seroconversion is defined as SRH area ≥25 mm2 for subjects who were seronegative at baseline [day 1 SRH area ≤3.997 mm2] or a significant increase [at least 50% increase] in SRH area for subjects who were seropositive at baseline [SRH area >3.997 mm2])
Percentage of subjects with geometric mean area ≥25 mm2 | day 43
Percentage of subjects achieving seroconversion | day 22
  Seroconversion is defined as HI ≥1:40 for subjects who were seronegative at baseline [day 1 HI titer <1:10] or a minimum 4-fold increase in HI titer for subjects who were seropositive at baseline [day 1 HI titer ≥1:10])
GMTs as determined by SRH | day 43 (3 weeks after the second vaccination)
  Serial radial haemolysis (SRH) assay: homologous antibody responses to aH5N1 vaccine 3 weeks after first and second vaccinations (day 22 and day 43) according to CHMP immunogenicity criteria in adult and elderly subjects who are healthy or with underlying medical condition
GMRs as determined by HI | day 22
Geometric mean titers (GMTs) as determined by HI | day 43 (3 weeks after the second vaccination)
  HI assay: homologous antibody responses to aH5N1 vaccine 3 weeks after first vaccination (day 22) according to CHMP immunogenicity criteria in adult and elderly subjects who are healthy or with underlying medical condition
Geometric mean titers (GMTs) as determined by HI | day 22 (3 weeks after the first vaccination)
  HI assay: homologous antibody responses to aH5N1 vaccine 3 weeks after first vaccination (day 22) according to CHMP immunogenicity criteria in adult and elderly subjects who are healthy or with underlying medical condition
GMRs as determined by SRH | day 43
Percentage of subjects with an HI titer ≥1:40 | day 1
Percentage of subjects with geometric mean area ≥25 mm2 | day 1
Percentage of subjects with geometric mean area ≥25 mm2 | day 22
Percentage of subjects achieving seroconversion | day 43
  Seroconversion is defined as SRH area ≥25 mm2 for subjects who were seronegative at baseline [day 1 SRH area ≤3.997 mm2] or a significant increase [at least 50% increase] in SRH area for subjects who were seropositive at baseline [SRH area >3.997 mm2])
GMTs as determined by SRH | day 1
  Serial radial haemolysis (SRH) assay: homologous antibody responses to aH5N1 vaccine 3 weeks after first and second vaccinations (day 22 and day 43) according to CHMP immunogenicity criteria in adult and elderly subjects who are healthy or with underlying medical condition
Geometric mean ratios (GMRs) as determined by SRH | day 43 (3 weeks after the second vaccination)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (6):
- Germany (6):
  - 001, Novartis Investigational Site, Berlin
  - 003, Novartis Investigational Site, Dresden
  - 005, Novartis Investigational Site, Hamburg
  - 006, Novartis Investigational Site, Magdeburg
  - 004, Novartis Investigational Site, Rostock
  - 002, Novartis Investigational Site, Würzburg

REFERENCES:
- [Background] Atmar RL, Keitel WA, Patel SM, Katz JM, She D, El Sahly H, Pompey J, Cate TR, Couch RB. Safety and immunogenicity of nonadjuvanted and MF59-adjuvanted influenza A/H9N2 vaccine preparations. Clin Infect Dis. 2006 Nov 1;43(9):1135-42. doi: 10.1086/508174. Epub 2006 Sep 25. PMID 17029131
- [Background] Banzhoff A, Gasparini R, Laghi-Pasini F, Staniscia T, Durando P, Montomoli E, Capecchi PL, di Giovanni P, Sticchi L, Gentile C, Hilbert A, Brauer V, Tilman S, Podda A. MF59-adjuvanted H5N1 vaccine induces immunologic memory and heterotypic antibody responses in non-elderly and elderly adults. PLoS One. 2009;4(2):e4384. doi: 10.1371/journal.pone.0004384. Epub 2009 Feb 6. PMID 19197383
- [Background] Podda A. The adjuvanted influenza vaccines with novel adjuvants: experience with the MF59-adjuvanted vaccine. Vaccine. 2001 Mar 21;19(17-19):2673-80. doi: 10.1016/s0264-410x(00)00499-0. PMID 11257408